CLINICAL TRIAL: NCT05445401
Title: A Pilot Study of Pre-rehabilitation in Neoadjuvant Patients With Gastric Cancer
Brief Title: Pre-rehabilitation in Neoadjuvant Patients With Gastric Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Quan Wang, Prof., The First Hospital of Jilin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STARS-GC06
Record Dates: First submitted 2022-06-23; First posted 2022-07-06 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Preoperative Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-rehabilitation group (Experimental): Triple pre-rehabilitation interventions of exercise, nutrition and psychology during the neoadjuvant period
  Interventions: Behavioral: Pre-rehabilitation
- Conventional group (Placebo Comparator): Conventional group
  Interventions: Behavioral: Standard medical care

INTERVENTIONS:
Behavioral: Pre-rehabilitation — Triple pre-rehabilitation interventions of exercise, nutrition and psychology
  Arms: Pre-rehabilitation group
Behavioral: Standard medical care — Traditional care
  Arms: Conventional group

SUMMARY:
In this study, patients with traditional neoadjuvant gastric cancer were used as controls to explore whether the triple pre-rehabilitation interventions of exercise, nutrition and psychology during the neoadjuvant period before surgery could improve the functional reserve of neoadjuvant gastric cancer patients and accelerate postoperative recovery.

DETAILED DESCRIPTION:
Internationally, pre-rehabilitation strategies have been widely used in surgery. Due to the late start of the concept of enhanced rehabilitation in my country, the research on pre-rehabilitation in my country is still in its infancy, and the research on pre-rehabilitation in gastric cancer is basically in a blank state. Domestic scholars have compared the rehabilitation of gastric cancer patients in the exercise-based pre-rehabilitation group and the postoperative rapid rehabilitation group, and found that the postoperative stress response, insulin resistance, and inflammatory response in the pre-rehabilitation group were lower than those in the conventional treatment group, and their nutritional status was improved. faster. The pre-rehabilitation model of comprehensive exercise, nutritional support and psychological intervention is rarely used in gastric cancer patients, and there is a lack of high-quality clinical data and related research.

Neoadjuvant chemotherapy and neoadjuvant chemotherapy combined with immunotherapy are the current research hotspots in locally advanced gastric cancer. The current research studies focus on tumor regression and prognosis and survival. However, the preoperative treatment cycle of neoadjuvant gastric cancer patients is long. If there is a lack of long-term and continuous effective management and guidance during the neoadjuvant therapy, it is very easy to lead to nutritional and nutritional deficiencies after neoadjuvant therapy. The poor physical condition makes the patient suffer from physical and psychological pain.

Therefore, we considered whether it is possible to carry out effective, convenient and economical rehabilitation training treatment for neoadjuvant gastric cancer patients before surgery, so as to prevent the occurrence of surgical risks and other complications in the preoperative stage, improve the functional reserve of neoadjuvant gastric cancer patients and respond to surgery. stimulated and accelerated postoperative recovery.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in clinical research, fully understand and inform this research and sign the Informed Consent Form (ICF), and are willing to follow and have the ability to complete all experimental procedures;
2. The age when signing the informed consent form is 18 to 65 years old, male or female;
3. Advanced gastric adenocarcinoma patients diagnosed with clinical stage II-III by CT, MRI, gastroscope and pathology (based on the 8th edition UICC/AJCC staging);
4. The function of major organs is normal;
5. No history of gastric cancer surgery, chemotherapy or immunotherapy;
6. Not accompanied by systemic infection requiring antibiotic treatment;
7. After general examination, it is planned to undergo neoadjuvant immunotherapy and neoadjuvant chemotherapy followed by surgery;
8. No contraindications related to CT and MRI examinations;
9. ECOG score of 0-2 points;

Exclusion Criteria:

1. The patient has a history of chemotherapy and immunotherapy in the past;
2. The patient cannot undergo CT or MRI scan, or has artifacts that cannot be assessed;
3. The patient refuses to participate in the study;
4. Patients who are going to undergo or have previously received organ or bone marrow transplantation;
5. The patient is pregnant, breastfeeding or unable to take appropriate contraceptive measures;
6. Patients with mental illness or related medical history, such as: the patient cannot understand the relevant requirements of this study;
7. Patients with human immunodeficiency virus (HIV) infection, active pulmonary tuberculosis or other severe, acute and chronic diseases that may increase the risk of participating in research and research drugs, and who are judged by the investigator to be unsuitable for participating in clinical research;
8. Other relevant factors are considered unsuitable for participating in the research by the researcher.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
6 minutes walking test | 1 month after surgery
  The maximum distance the patient can walk on an unimpeded hard surface in six minutes.
Scored Patient-Generated Subjective Global Assessment score | 1 month after surgery
  Scored Patient-Generated Subjective Global Assessment(PG-SGA), PG-SGA consists of two parts: patient self-assessment and medical staff assessment. The specific contents include body weight, food intake, symptoms, activity and physical function, the relationship between disease and nutritional needs, metabolic needs, Physical examination and other 7 aspects, the first 4 aspects are evaluated by the patients themselves, and the last 3 aspects are evaluated by the medical staff. The overall evaluation includes qualitative evaluation and quantitative evaluation. Higher scores mean a worse outcome.
DMSM score | 1 month after surgery
  Distress Management Screening Measure(DMSM）, is an assessment tool recommended by the US National Comprehensive Cancer Network for screening the level and possible causes of psychological pain. The DMSM questionnaire consists of two parts: the first part is the Psychological Distress Thermometer (DT). The second part is the problem list (PL), which contains 36 factors.Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Quality of life score QLQ-C30 | 3 month after surgery
  Assessed using the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaires (QLQ-C30 ).
Quality of life score QLQ-STO22 | 3 month after surgery
  Assessed using the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaires ( QLQ-STO22).
Postoperative skeletal muscle index of the third lumbar spine plane. | 3 month after surgery
  Grip strength (Kg).
The rate of weight loss (≥10%) . | 3 month after surgery
  The rate of weight loss (≥10%) .
The incidence of sarcopenia. | 3 month after surgery
  The incidence of sarcopenia.
The ratio of actual ONS to recommended ONS. | 3 month after surgery
  The ratio of actual ONS to recommended ONS.
Albumin | 3 month after surgery
  Laboratory test: albumin （g/L）
Hemoglobin | 3 month after surgery
  Laboratory test: hemoglobin (g/L)
Prealbumin. | 3 month after surgery
  Laboratory test: prealbumin (g/L)
Incidence of adverse reactions during neoadjuvant therapy. | 1 month after surgery
  Incidence of adverse reactions during neoadjuvant therapy.
Completion rate of neoadjuvant therapy for gastric cancer | 1 month after surgery
  Number of completed courses/number of regimen courses
Surgery rate after neoadjuvant therapy for gastric cancer. | 1 month after surgery
  Surgery rate after neoadjuvant therapy for gastric cancer.
TRG grading after neoadjuvant therapy for gastric cancer. | 1 month after surgery
  TRG grading after neoadjuvant therapy for gastric cancer.
R0 resection rate | 1 month after surgery
  R0 resection rate
Postoperative complication rate of grade IIIa or above. | 3 month after surgery
  Postoperative complication rate of grade IIIa or above.

CONTACTS AND LOCATIONS:
Overall Officials: Quan Wang, Principal Investigator — The First Hospital of Jilin University

IPD SHARING:
Plan to Share IPD: No